CLINICAL TRIAL: NCT00508703
Title: Pilot Study of Intensity Modulated Radiotherapy (IMRT) to Pelvis Post-Hysterectomy With Analysis of Clinical Target Volume Motion and Relation to Position and Volume of Bladder and Rectum During Course of Radiotherapy for Use in Optimization of Margin Size
Brief Title: Intensity Modulated Radiotherapy (IMRT) for the Pelvis Post-Hysterectomy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID03-0047
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Uterine Cancer; Cervical Cancer; Endometrial Cancer
Keywords: Uterine Cancer; Cervical Cancer; Endometrial Cancer; Intensity Modulated Radiotherapy; IMRT; Computed Tomography; CT; CT Scan
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT Scan + IMRT Radiation Therapy
  Interventions: Radiation: Intensity Modulated Radiotherapy (IMRT); Procedure: CT Scan

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy (IMRT) — Dose of 45Gy
Procedure: CT Scan — CT Scans: Twice a week during the 5 weeks of radiation treatment.
  Other Names: Computed Tomography

SUMMARY:
The goal of this clinical research study is to use CT scans to find any changes in position of the vagina and pelvic lymph node areas during the course of IMRT radiation therapy. Treatment can then be adjusted in order to "spare" as much normal tissue as possible during radiation therapy. Another goal is to study the side effects of IMRT radiation therapy.

DETAILED DESCRIPTION:
The standard radiotherapy technique for delivering radiation therapy to the pelvis following a hysterectomy involves a technique which also causes a large amount of normal tissue to receive radiation. This can cause both early and late side effects, which may be severe. The new technique of intensity modulated radiotherapy (IMRT) has been used to help spare normal tissue, especially tissue of the small bowel. This is an advanced new technology that delivers the high-dose of radiation to the target area but avoids the normal tissue. Using CT scans, the target is outlined by the doctors before treatment. However, sometimes organs in the pelvis move throughout the course of treatment. Using CT scans during treatment and re-outlining the target may help to deliver more radiation to the cancer tissues and less to the surrounding normal areas.

During the study, you will have additional CT scans that will be performed on a special scanner in the radiation treatment room. You also will have additional CT scans twice a week during the 5 weeks of radiation treatment. The first 12 participants enrolled will receive the standard radiation therapy taking into account the maximum possible movements of the bladder. No adjustments will be made according to the results of the additional CT scans. The next 12 participants may have their radiation therapy adjusted according to the CT scans in an effort to target less of the normal tissue without missing cancer tissue. To reduce movement of your bladder due to different amounts of fluid in your bladder, you will be asked to drink 3 glasses of water before treatment and to come for treatment with a full bladder.

The volumes of your bladder and rectum will also be studied, and any side effects of the treatment will be recorded. You will be asked to fill out a short questionnaire about the side effects of your treatment 3 times per week during treatment. It should take around 5 minutes to complete the questionnaire.

Patients will be followed for at least 2 years. (Every 3 months for 1 year and 4 months for second year according to usual clinic practice.)

This is an investigational study. IMRT radiation therapy is an approved method of treating some types of cancer. However, adjusting the radiation treatment according to the movement of the internal organs is investigational. Initial CT scans for treatment planning are part of standard treatment. Up to 24 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been treated with a hysterectomy for carcinoma of the uterine cervix or endometrium who require post-operative radiation or chemoradiation therapy because of positive pelvic lymph nodes or other high-risk local findings.
2. Patients must have no evidence of metastatic disease outside of the pelvis.
3. Patients must have a Karnofsky Performance Status of >60.
4. The patient must be able to understand the protocol and sign a study-specific informed consent. .

Exclusion Criteria:

1. Karnofsky Performance Status < 60.
2. Patients with para-aortic nodal disease or who require extended field radiotherapy beyond the pelvis.
3. Obese patients who exceed the size limits of hte treatment table or CT scanner.
4. Mental status changes or bladder control problems that make the patient unable to comply with bladder-filling instructions.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women treated with a hysterectomy for carcinoma of the uterine cervix or endometrium who require post-operative radiation or chemoradiation therapy because of positive pelvic lymph nodes or other high-risk local findings.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2003-03-05 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Maximum variations in position of the vagina and lymph node regions caused by bladder filling and emptying | 2 Years (every 3 months for first year and 4 months for second year)

SECONDARY OUTCOMES:
Day-to-day variations in position of vaginal vault and pelvic lymph node regions | During a 5-week course of intensity modulated pelvic radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J. Eifel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org